CLINICAL TRIAL: NCT01024478
Title: Contrast-Enhanced Whole-Heart Coronary Magnetic Resonance Angiography at 3.0-T: A Multicenter Trial
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Fujian Medical University Union Hospital (Other); Air Force Military Medical University, China (Other); Huazhong University of Science and Technology (Other); Nanjing Medical University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Henan Provincial People's Hospital (Other); Fudan University (Other)
Responsible Party: Li,kuncheng, Radiology department of Xuanwu Hospital
Other Study IDs: CapitalMedicalU
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery; Magnetic Resonance Angiography; Coronary Artery disease; Multicenter Trial; Cardiac MRI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The multicenter study evaluates the diagnostic performance of 3.0 T contrast-enhanced whole-heart coronary MRA in patients with suspected coronary artery disease.

DETAILED DESCRIPTION:
This is a multicenter trial evaluated the diagnostic ability of 3.0 T contrast-enhanced whole-heart coronary MRA to detect significant coronary artery stenosis among patients with suspected CAD.

A total of 272 patients will be prospectively enrolled from 8 cities in China.

ELIGIBILITY:
Inclusion Criteria:

* Suspected CAD, scheduled for DSA
* Sinus rhythm

Exclusion Criteria:

* Contraindications to MR examination: pacemaker, intraauricular implants, intracranial clips, thoracotomy, claustrophobia, orthopnea
* Acute coronary syndrome
* Atria fibrillation
* Coronary stents
* Bypass grafts
* Renal insufficiency (estimated glomerular filtration rate assessed by creatinine clearance <60 ml/min/1.73 m2)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive eligible patients scheduled to undergo conventional coronary angiography.
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: kuncheng li, M.D., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Radiology Department of Xuanwu Hopital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Yang Q, Li K, Liu X, Bi X, Liu Z, An J, Zhang A, Jerecic R, Li D. Contrast-enhanced whole-heart coronary magnetic resonance angiography at 3.0-T: a comparative study with X-ray angiography in a single center. J Am Coll Cardiol. 2009 Jun 30;54(1):69-76. doi: 10.1016/j.jacc.2009.03.016. PMID 19555843